CLINICAL TRIAL: NCT07281703
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HY8931 Following Single Intravenous and Multiple Subcutaneous Doses in Healthy Participants
Brief Title: Evaluation of the Safety, Tolerability and Pharmacokinetics of HY8931 in Healthy Adult Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Newsoara Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Newsoara HYK Biopharmaceutical (Shanghai) Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HY8931-01-01
Record Dates: First submitted 2025-11-19; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HY8931 (Experimental): It's an injection solution. SAD part for intravenous dosing in 6 cohorts, including 10mg, 30mg, 60mg, 120mg, 240mg and 360mg with only one administration on Day 1 of each cohort. SAD part for subcutaneous dosing in 120mg cohort with only one administration on Day 1; MAD part for subcutaneous dosing in 3 cohorts, including 120mg, 240mg, 360mg with two administrations on Day 1 and Day 30 of each cohort.
  Interventions: Biological: HY8931
- placebo (Placebo Comparator): It's same injection solution just without active ingredient compared with HY8931. SAD part for intravenous dosing in 6 cohorts, including 10mg, 30mg, 60mg, 120mg, 240mg and 360mg with only one administration on Day 1 of each cohort. SAD part for subcutaneous dosing in 120mg cohort with only one administration on Day 1; MAD part for subcutaneous dosing in 3 cohorts, including 120mg, 240mg, 360mg with two administrations on Day 1 and Day 30 of each cohort.
  Interventions: Other: Placebo Control

INTERVENTIONS:
Biological: HY8931 — HY8931 is an injection solution with 125mg/ml per vial. SAD part for intravenous dosing in 6 cohorts, including 10mg, 30mg, 60mg, 120mg, 240mg and 360mg and for subcutaneous dosing in 1 cohort of 120mg with only one administration on Day 1 of each cohort. MAD part for subcutaneous dosing in 3 cohorts, including 120mg, 240mg and 360mg with two administrations on Day 1 and Day 30 of each cohort.
  Arms: HY8931
Other: Placebo Control — A vial with 1ml injection solution contain same ingredient except HY8931 compared with HY8931 solution.
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to learn the safety, tolerability and pharmacokinetics of single and multiple doses of HY8931 in healthy adult participants. The main questions it aims to answer are:

* How is the safety and tolerability following administration of single and multiple doses of HY8931 in healthy adult participants?
* What is the PK character of HY8931 following administration of single and multiple doses of HY8931 in healthy adult participants?

Researchers will compare HY8931 to a placebo (a look-alike substance that contains no drug) to see if HY8931 is safe and well tolerated.

Participants will take HY8931 or a placebo once or twice in single dose group or multiple dose group. And will be follow-up until Day 90.

DETAILED DESCRIPTION:
The rationale of the study is by simultaneously targeting TL1A and IL-23p19, HY8931 as an investigational bispecific antibody, presents a novel and promising therapeutic strategy. It has the potential to disrupt multiple pathogenic pathways in IBD, effectively breaking the vicious cycle of inflammation. Pre-clinical studies have demonstrated that the dual inhibition of these cytokines can effectively reduce eosinophilic inflammation, airway hyperresponsiveness, and tissue remodeling in animal models. This approach holds the potential to not only alleviate acute symptoms but also modify the disease course, offering a more comprehensive and effective treatment strategy for patients suffering from these debilitating respiratory conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 18 to 45 years of age, inclusive, at the time of signing the informed consent.
2. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital sign and 12-lead ECG.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. BMI of 18 to 32 kg/m2; and a total body weight >50 kg.
5. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Positive hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody or positive testing for HIV or syphilis at the screening visit.
3. History of allergic or anaphylactic reaction to a therapeutic drug.
4. History of recent active infections within 28 days prior to the screening visit.
5. Participants with a fever within 48 hours prior to dosing.
6. Positive QFT-G test.
7. History of recurrent bacterial infection (>3 per year) or recurrent HSV infection.
8. The medications as listed in section 6.9.2 are exclusionary, all other medications and supplements allowed at investigator discretion. (Refer to Section 6.9 Prior and Concomitant Therapy for additional details).
9. Recent exposure to live vaccines within 28 days of the screening visit or plan to receive live vaccination during the trial.
10. Known exposure to anti-TL1A or IL23 or any type of anti-TL1A or anti-IL23 therapy.
11. Previous administration with an investigational drug within 90 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
12. A positive urine drug test.
13. A positive pregnancy test.
14. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
15. Baseline 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTc interval>450 msec, complete LBBB, signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second or third-degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected- using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer interpreted-ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
16. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific-laboratory and confirmed by a single repeat test, if deemed necessary:

    * AST or ALT level >1.5 × ULN;
    * Total bilirubin level >1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN;
17. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week for male, 10 units per week for female (1 unit = 240 mL beer, 30 mL of 40% spirit or 90 mL of wine). And participants with >5 cigarettes per week intake.
18. Blood donation (excluding plasma donations) of approximately 500 mL or more within 30 days prior to dosing.
19. History of sensitivity to heparin or heparin -induced thrombocytopenia
20. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
21. Investigator site staff or The sponsor employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From signing informed consent form to the end of study at Day 90.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | From Day1 predose to Day 90.
Area under the plasma concentration versus time curve (AUC) | From Day1 predose to Day 90.
Time to maximum concentration (Tmax) | From Day1 predose to Day 90.
Plasma half-life time (T1/2) | From Day1 predose to Day 90.

CONTACTS AND LOCATIONS:
Overall Officials: Weifen Zhou, Dr., Study Director — Newsoara Biopharma Co., Ltd.
Locations (1):
- Q-Pharm Pty Ltd., Brisbane, Australia

IPD SHARING:
Plan to Share IPD: No